CLINICAL TRIAL: NCT01508975
Title: Satiety Response of White and Brown Rice Compared to Glucose Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 11028E03765
Record Dates: First submitted 2012-01-09; First posted 2012-01-12 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Food Selection
Keywords: satiety; obesity; food intake
MeSH Terms: conditions — Food Preferences; Obesity | interventions — Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- white rice (Experimental): White rice
  Interventions: Other: White Rice, Brown Rice, Glucose
- Brown rice (Experimental): Brown Rice
  Interventions: Other: White Rice, Brown Rice, Glucose
- Glucose (Experimental): Glucose
  Interventions: Other: White Rice, Brown Rice, Glucose

INTERVENTIONS:
Other: White Rice, Brown Rice, Glucose — white rice, brown rice, glucose

SUMMARY:
The investigators hypothesize that consumption of either white or brown rice will be more satiating than glucose control.

DETAILED DESCRIPTION:
This study is an acute, randomized, repeated measures design with 20 subjects. Subjects will consume 3 test breakfasts, white rice, brown rice, or glucose control, each containing 400 calories. Treatments will be one week apart. After consumption of the controlled breakfast, subjects will complete visual analogue scales (VAS) for satiety response. Additionally, they will consume a pizza lunch and record food intake for the next 24 hours. Breath gas samples will be collected to estimate fermentation of fiber in the large intestine. Also, subjective data on gastrointestinal tolerance will be collected.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects

Exclusion Criteria:

* inability to consume rice for breakfast

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Satiety | 4 hours following breakfast
  Visual analogue scales (subjective measurements)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Slavin, PhD, Principal Investigator — University of Minnesota
Locations (1):
- Department of Food Science and Nutrition, Saint Paul, Minnesota, United States